CLINICAL TRIAL: NCT00445367
Title: Large-scale, Multi-disciplinary Sample and Data Repository for Multiple Sclerosis and Related Demyelinating Diseases
Brief Title: Biobank For MS And Other Demyelinating Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Accelerated Cure Project for Multiple Sclerosis (Other)
Responsible Party: Sponsor
Other Study IDs: ACP-001
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Transverse Myelitis; Neuromyelitis Optica; Acute Disseminated Encephalomyelitis; Optic Neuritis
Keywords: Multiple Sclerosis; Clinically Isolated Syndrome; Transverse Myelitis; Neuromyelitis Optica; Acute Disseminated Encephalomyelitis; Optic Neuritis; Repository; Biobank
MeSH Terms: conditions — Multiple Sclerosis; Myelitis, Transverse; Neuromyelitis Optica; Encephalomyelitis, Acute Disseminated; Optic Neuritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
- Control

SUMMARY:
To establish a large, longitudinal collection of high quality samples and data from subjects with MS, selected other demyelinating diseases (Transverse Myelitis (TM), Neuromyelitis Optica (NMO) or Devic's, Acute Disseminated Encephalomyelitis (ADEM), and Optic Neuritis (ON)), and related and unrelated unaffected controls. Samples and data will be available as a shared resource to scientists researching the causes, sub-types, and biomarkers of MS and related demyelinating diseases.

ELIGIBILITY:
Inclusion Criteria:

* age 18+ able to give informed consent or individuals younger than 18 with parental permission and able to give assent
* willing to provide up to 110 ml (50 ml for < 18 years old) of blood via venipuncture
* experienced at least one CNS demyelinating event characteristic of MS, TM, NMO, ADEM, or ON

Exclusion Criteria:

* history of blood borne pathogens
* allogeneic bone marrow transplant
* clinical or radiological evidence of stroke, meningitis, or other well characterized diseases of the nervous system (with the exception of MS, TM, NMO, ADEM, or ON).
* weight less than 37 pounds

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with MS, selected other demyelinating diseases (Transverse Myelitis (TM), Neuromyelitis Optica (NMO) or Devic's, Acute Disseminated Encephalomyelitis (ADEM), and Optic Neuritis (ON)), and related and unrelated unaffected controls.
Sampling Method: Non-Probability Sample
Enrollment: 3226 (Actual)
Dates: Start 2006-05; Primary Completion 2030-10 (Estimated); Study Completion 2036-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, M.D., M.H.S., Principal Investigator — University of Texas
Locations (10):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Stanford University, Stanford, California
  - The Rocky Mountain MS Center at Anschutz Medical Campus at UC Denver, Aurora, Colorado
  - Shepherd Center, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Multiple Sclerosis Research Center of New York, New York, New York
  - The Ohio State University, Columbus, Ohio
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- See also: Accelerated Cure Project MS Repository Overview — https://www.acceleratedcure.org/research/acp-repository/